CLINICAL TRIAL: NCT06846801
Title: Evaluation of the Outcomes of Endoscopic Balloon Dilation Under X-DR Portable X-ray System Guidance in the Treatment of Pharyngo-oesphageal Strictures
Brief Title: Balloon Dilation Under Portable X-ray System in the Treatment of Pharyngo-oesphageal Strictures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Elrabie Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mohammed Elrabie Ahmed, Mahmoud Ibrahim Yousef, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-1-9PD
Record Dates: First submitted 2025-02-07; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pharyngo-oesphageal Strictures

STUDY DESIGN:
Intervention Model Description: 20 patients who will attend to Sohag university hospital and will be diagnosed to have oesophageal strictures regardless of the age of the patient (previously dilated strictures, neoplastic strictures and post-irradiation strictures will be excluded from the study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- one (Experimental): 20 patients who will attend to Sohag university hospital and will be diagnosed to have oesophageal strictures regardless of the age of the patient (previously dilated strictures, neoplastic strictures and post-irradiation strictures will be excluded from the study).
  Interventions: Procedure: Balloon Dilation Under Portable X-ray System

INTERVENTIONS:
Procedure: Balloon Dilation Under Portable X-ray System — * All the esophageal dilation procedures will be performed using rigid hypopharyngoscope and / or oesophagoscope with endotracheal intubation under general anesthesia by experienced surgical and anesthesia team.
  * The rigid hypopharyngoscope / oesophagoscope (Storz, germany) will be introduced through the mouth to whole through examination to localize the site of the stenosis then a contrast material will be injected via the endoscope and picture taken with X-DR portable x-ray system.
  * After that a guide wire 0.035mm will be passed through the endoscope till the stomach. The guide wire site will be confirmed by with X-DR portable x-ray system and then a suitable size balloon catheter will be passed over the guide wire (Boston Scientific, Cork, Ireland), then the balloon catheter will be advanced through the stricture confirmed by taking a photo by the x-ray system. The balloon will be inflated with radiopaque contrast solution using EncoreTM 26 inflation device.

SUMMARY:
The aim of our study is to evaluate the outcomes (efficacy and safety) and to present our experience in X-DR portable x-ray system guided endoscopic balloon dilatation in the treatment of pharyngo-oesophageal strictures as an alternative procedure to the videofluroscopic guided maneuver.

DETAILED DESCRIPTION:
The study will include 20 patients who will attend to Sohag university hospital and will be diagnosed to have oesophageal strictures regardless of the age of the patient (previously dilated strictures, neoplastic strictures and post-irradiation strictures will be excluded from the study).

* The diagnosis of oesophageal stricture and need of patients for dilatation will be determined according to symptoms such as dysphagia clinical score (simplified dysphagia severity rating scale mentioned previously), decreased tolerance depending on the consistency and caliber of the food pieces, water soluble upper gastrointestinal contrast radiographies, and sometimes the need for flexible upper GIT endoscopy.
* All the esophageal dilation procedures will be performed using rigid hypopharyngoscope and / or oesophagoscope with endotracheal intubation under general anesthesia by experienced surgical and anesthesia team.
* The rigid hypopharyngoscope / oesophagoscope (Storz, germany) will be introduced through the mouth to whole through examination to localize the site of the stenosis then a contrast material will be injected via the endoscope and picture taken with X-DR portable x-ray system.
* After that a guide wire 0.035mm will be passed through the endoscope till the stomach. The guide wire site will be confirmed by with X-DR portable x-ray system and then a suitable size balloon catheter will be passed over the guide wire (Boston Scientific, Cork, Ireland), then the balloon catheter will be advanced through the stricture confirmed by taking a photo by the x-ray system. The balloon will be inflated with radiopaque contrast solution using EncoreTM 26 inflation device. Before inflation, correct placement of the deflated balloon will be checked with X-DR portable x-ray system.
* The length of the balloon will be -35.5 cm, and the diameters range from 6 to 20 mm and will be translucent in color. The balloon will be inflated up to 4-10 atm pressure and kept inflated for 3 to 5 min.
* After confirming the persistence of the ''waist'' and that it will be both endoscopically and image guided safe, the diameter of the balloon will be increased.
* Appropriate balloon catheter size will be determined by the surgeon by evaluating the patient's age, body weight, the severity of the esophageal stricture determined on the barium image.
* After deflation and removal of balloon, the contrast material will be injected through the rigid endoscope and an image by the portable system will be taken as a post dilatation check test for the possibility of oesophageal perforation.
* Antibiotic prophylaxis and proton pump inhibitors will be routinely prescribed unless there will be any complications. All patients will undergo chest X-ray 12 hours after the procedure. If no pathological finding is detected in the patients' examination and chest X-ray, the patients will be encouraged to start feeding orally with gradual introduction of clear fluids, soft food then solids and discharged 3-4 hours after that. Upper GI contrast study will not performed routinely in asymptomatic patients. Patients with severe strictures will be called back after 4-6 weeks. Symptom monitoring will be recommended for patients with mild strictures and no need for dilation for more than 3 months.

  * All of the patients' demographic features, primary diagnosis, additional diseases, level of stricture, type of stricture (simple, complex), total number of dilations, balloon sizes used in the first and last dilation, time between dilations, complications due to the procedure, gastrostomy opening, need for additional surgical procedure, therapeutic agent injection, trial of C-mac, preoperative upper GI contrast radiographies, time spent without the need for dilation, and the follow-up time will be recorded and statistically analyzed using the suitable statistical tests.
  * Efficacy will be measured by improvements in symptoms (e.g., dysphagia scores, quality of life), the number of dilatation sessions required, and overall long-term outcomes.
  * Safety will involve tracking complications, such as perforations, bleeding, and other adverse events

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed to have oesophageal strictures with clinical and radiological investigation regardless of the age of the patient

Exclusion Criteria:

* previously dilated strictures
* neoplastic strictures
* Post-irradiation strictures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Treatmet of pharyngo-oesphageal strictures | 6 months
  improvements in dysphgia scores

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mohammed Elrabie Ahmed, Sohag
  - Sohag University, Sohag

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Standards of Practice Committee; Egan JV, Baron TH, Adler DG, Davila R, Faigel DO, Gan SL, Hirota WK, Leighton JA, Lichtenstein D, Qureshi WA, Rajan E, Shen B, Zuckerman MJ, VanGuilder T, Fanelli RD. Esophageal dilation. Gastrointest Endosc. 2006 May;63(6):755-60. doi: 10.1016/j.gie.2006.02.031. No abstract available. PMID 16650533
- [Background] Azizkhan RG, Stehr W, Cohen AP, Wittkugel E, Farrell MK, Lucky AW, Hammelman BD, Johnson ND, Racadio JM. Esophageal strictures in children with recessive dystrophic epidermolysis bullosa: an 11-year experience with fluoroscopically guided balloon dilatation. J Pediatr Surg. 2006 Jan;41(1):55-60; discussion 55-60. doi: 10.1016/j.jpedsurg.2005.10.007. PMID 16410108